CLINICAL TRIAL: NCT04769817
Title: Prostate Cancer Theranostics and Imaging Centre of Excellence (ProsTIC) Prospective Patient Registry of Men Treated With PSMA Theranostics
Brief Title: ProsTIC Registry of Men Treated With PSMA Theranostics
Status: Recruiting | Type: Observational
Sponsor: Peter MacCallum Cancer Centre, Australia (Other)
Responsible Party: Sponsor
Other Study IDs: PMC 20/164
Record Dates: First submitted 2020-09-06; First posted 2021-02-25 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-04

CONDITIONS: Prostate Cancer; Metastatic Castration-resistant Prostate Cancer
Keywords: Prostate Cancer; Metastatic Castration-resistant Prostate Cancer; Theranostic; 177Lu-PSMA; Radionuclide Therapy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Biospecimen Retention: Samples With DNA — Prognostic and predictive biomarkers associated with treatment outcome and response will be assessed. This will include any of the following:
  i. Circulating tumour deoxyribonucleic acid (DNA) ± tumour tissue (DNA repair genes, tumour suppressor genes, androgen receptor); and ii. Whole blood ribonucleic acid (RNA) (androgen receptor splice variants, TMPRSS2:ERG fusion) iii. Blood or histopathology parameters
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: 177Lu-PSMA — Lu-PSMA will be administered as a standard-of-care procedure following assessment of suitability by a nuclear medicine physician and managed in close collaboration with the patient's medical oncologist.

SUMMARY:
This is a descriptive, observational, prospective, open-ended, registry utilising electronic data capture to collect information on the outcomes of men treated with prostate specific-membrane antigen (PSMA) theranostics.

DETAILED DESCRIPTION:
The aim of the registry is to collect data of men with pre-treated metastatic castration-resistant prostate cancer (mCRPC) receiving Lutetium 177 (177Lu)-PSMA outside of a clinical trial to assess "real world" anti-tumour utility. The primary objective is to assess prostate specific antigen (PSA) response rate to 177Lu-PSMA in men with mCRPC.

Patients with mCRPC who have have progression or intolerance on a novel anti-androgen targeted agent (abiraterone and/or enzalutamide and/or apalutamide) will be eligible for the study.

The investigators intend to evaluate the safety of 177Lu-PSMA, in addition to determining patient PSA progression-free survival (PFS), objective radiographic response rates and overall survival (OS). Health-related quality of life (QoL) and pain will also be observed. Additional objectives are to identify biomarkers and assess the relationship between PSMA and F-fluorodeoxyglucose (FDG) Positron Emission Tomography-Computed Tomography (PET/CT) parameters associated with clinical outcomes.

ELIGIBILITY:
Inclusion criteria:

1. Diagnosis of mCRPC
2. Progression or intolerance on a novel anti-androgen therapy (e.g. abiraterone, enzalutamide, apalutamide or darolutamide)
3. Prior therapy with at least one taxane cytotoxic (these agents may have been received upfront for metastatic hormone-sensitive prostate cancer) or the patient is symptomatic and assessed as unfit for chemotherapy
4. Referred to nuclear medicine and being considered for Lu-PSMA therapy according to institutional procedure guidelines

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Men with metastatic castration-resistant prostate cancer (mCRPC).
Study Population: Men with mCRPC who have progressed after novel anti-androgen therapy and taxane chemotherapy (unless unfit and symptomatic).
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
PSA-RR | From baseline through to progression or death until registry completion (approx. 5 years).
  Prostate specific antigen-response rate (PSA-RR) defined as the proportion of participants with a PSA reduction of ≥ 50 percent from baseline.

SECONDARY OUTCOMES:
Number of participants with Adverse Events (AE) and Serious Adverse Events (SAE) measured using National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0 | From date of treatment to 12 weeks after completing study treatment.
  Safety of the combination will be measured by selected AEs and SAEs; only grade 3 or greater AEs related to 177Lu-PSMA with the exception of lymphopenia and fatigue or any grade 1-2 AEs that have not previously been reported with 177Lu-PSMA
Radiographic progression-free survival (rPFS) | From date of treatment through to progression or death until registry completion (approx. 5 years).
  rPFS is defined as the time from treatment initiation to the first date of documented radiographic progression using conventional imaging or death due to any cause, whichever occurs first. The radiographic progression will be assessed by the investigator per response evaluation criteria in solid tumors (RECIST1.1) for soft tissue and prostate cancer working group three (PCWG3) for bone lesions.
PSA progression free survival (PSA-PFS) | From date of treatment through to progression or death until registry completion (approx. 5 years).
  PSA-PFS is defined as the time from treatment initiation to the date of PSA progression per PCWG3 or death due to any cause, whichever occurs first. The date of PSA progression is the date that an increase of 25% or more and an absolute increase of 2ng/mL or more from the nadir is documented. For patients who have an initial PSA decline during treatment, this must be confirmed by a second value 3 or more weeks later.
Overall survival (OS) | From date of treatment, up until 18 months after the last patient commences treatment.
  OS is defined as the time from treatment initiation to the date of death due to any cause.
EORTC QLQ-C30 | From baseline through to progression or death until registry completion (approx. 5 years).
  The European Organization for Research and Treatment of Cancer core quality of life questionnaire (EORTC QLQ-C30) includes five functional scales (physical, role, cognitive, emotional, and social), three symptom scales (fatigue, pain, and nausea and vomiting), and a global health and quality-of-life scale. The remaining single items assess additional symptoms commonly reported by cancer patients (dyspnoea, appetite loss, sleep disturbance, constipation, and diarrhoea), as well as the perceived financial impact of the disease and treatment.
  All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. Thus a high score for a functional scale represents a high/healthy level of functioning, a high score for the global health status/QoL represents a high QoL, but a high score for a symptom scale/item represents a high level of symptomatology/problems.
PPI | From baseline through to progression or death until registry completion (approx. 5 years).
  Pain is measured using the McGill-Melzack Present Pain Intensity scale (PPI) Pain Response is defined for patients with a baseline PPI score of ≥2 or a baseline analgesic score of ≥10 points, as: (i) a PPI score reduction of ≥2 points from baseline with no increase in analgesic score; and/or, (ii) a decrease of ≥ 50 percent in analgesic score with no increase PPI.

OTHER OUTCOMES:
Prognostic and predictive value of baseline PET/CT | Baseline PSMA and FDG PET/CT within 3 months of 177Lu-PSMA therapy.
  PET-derived parameters including molecular tumour volume parameters (volume, SUVmax, SUVmean) and other parameters including radiomics from PET, CT, post therapy SPECT/CT or bone scans using data-characterisation algorithms will be assessed
Prognostic value of 12 week restaging PSMA and FDG PET/CT | 12 weeks after first cycle of 177Lu-PSMA therapy.
  PET-derived parameters including molecular tumour volume parameters (volume, SUVmax, SUVmean) and other parameters including radiomics from PET, CT, post therapy SPECT/CT or bone scans using data-characterisation algorithms will be assessed
Histopathology parameters | At baseline, 12 weeks post treatment and date of progression.
  Histological grading of adenocarcinoma of the prostate (obtained via biopsy) using the International Society of Urological Pathology (ISUP) modified Gleason Grades. The cells identified are given a grade number from 1 to 5, depending on the abnormality of the cells, 1 being the lowest, 5 the highest. The grades of the two most common patterns are added together to give a score from 2 to 10. The higher the score, the more aggressive and fast-growing the cancer.
Tumour DNA ± tumour tissue | At baseline, 12 weeks post treatment and date of progression.
  Measurement of prognostic and predictive biomarkers (Circulating tumour deoxyribonucleic acid (DNA) ± tumour tissue (DNA repair genes, tumour suppressor genes, androgen receptor) associated with treatment outcome and response
Whole blood RNA (androgen receptor splice variants) | At baseline, 12 weeks post treatment and date of progression.
  Measurement of prognostic and predictive biomarkers. Alterations in whole blood ribonucleic acid (RNA) androgen receptor splice variants
Whole blood RNA (TMPRSS2:ERG fusion gene) | At baseline, 12 weeks post treatment and date of progression.
  Measurement of prognostic and predictive biomarkers. Alterations in whole blood ribonucleic acid (RNA) TMPRSS2:ERG fusion

CONTACTS AND LOCATIONS:
Locations (1):
- Peter MacCallum Cancer Centre, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No